CLINICAL TRIAL: NCT00070304
Title: A Phase II Study Of Weekly Gemcitabine And Vinorelbine In Children With Recurrent Or Refractory Hodgkin's Disease
Brief Title: Gemcitabine and Vinorelbine in Treating Young Patients With Recurrent or Refractory Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AHOD0321; CDR0000331915 (Other: Clinical Trials.gov); COG-AHOD0321 (Other: Children's Oncology Group)
Record Dates: First submitted 2003-10-03; First posted 2003-10-07 (Estimated); Last update posted 2013-07-26 (Estimated); Status verified 2013-07

CONDITIONS: Lymphoma
Keywords: recurrent/refractory childhood Hodgkin lymphoma; childhood lymphocyte predominant Hodgkin lymphoma; childhood lymphocyte depletion Hodgkin lymphoma; childhood nodular sclerosis Hodgkin lymphoma; childhood mixed cellularity Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Recurrence; Hodgkin Disease | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; Gemcitabine; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Patients receive vinorelbine tartrate IV over 6-10 minutes and gemcitabine hydrochloride IV over 100 minutes on days 1 and 8. Patients also receive filgrastim (G-CSF) subcutaneously daily beginning on day 9 and continuing for at least 7 days and until blood counts recover. Treatment repeats every 21 days for at least 2 courses in the absence of disease progression or unacceptable toxicity. Patients with responding disease after 2 courses may proceed directly to stem cell transplantation off study OR receive 2 additional courses. Patients with stable disease after 2 courses receive at least 2 additional courses. Patients with continued stable or responding disease (with no disease progression) after 4 courses may continue to receive study treatment for up to 1 year or discontinue study for alternative therapy at the discretion of the treating physician.
  Interventions: Biological: filgrastim; Drug: gemcitabine hydrochloride; Drug: vinorelbine tartrate

INTERVENTIONS:
Biological: filgrastim — Given by mouth or IV, 5 micrograms/kg/dose (up to 10 micrograms/kg/dose) daily starting on day 9 for a minimum of 7 days and until the ANC is greater to or equal to 1,500/uL.
  Other Names: Granulocyte Colony-Stimulating Factor; r-metHuG-CSF; G-CSF; Neupogen; NSC # 614629
Drug: gemcitabine hydrochloride — Given IV over 100 minutes dose 1000 mg/m2/dose in 500 ml NS on days 1 and 8
  Other Names: Gemzar; NSC #613327
Drug: vinorelbine tartrate — Given IV over 6-10 minutes (central venous catheter). Dose 25 mg/m2/dose on days 1 and 8
  Other Names: Navelbine; NSC #608210

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine and vinorelbine, use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving gemcitabine together with vinorelbine works in treating young patients with recurrent or refractory Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate of pediatric patients with recurrent or refractory Hodgkin's lymphoma treated with gemcitabine and vinorelbine.
* Determine the toxicity of this regimen in these patients.

OUTLINE: This is a nonrandomized, multicenter study.

Patients receive vinorelbine IV over 6-10 minutes and gemcitabine IV over 100 minutes on days 1 and 8. Patients also receive filgrastim (G-CSF) subcutaneously daily beginning on day 9 and continuing for at least 7 days and until blood counts recover. Treatment repeats every 21 days for at least 2 courses in the absence of disease progression or unacceptable toxicity. Patients with responding disease after 2 courses may proceed directly to stem cell transplantation off study OR receive 2 additional courses. Patients with stable disease after 2 courses receive at least 2 additional courses. Patients with continued stable or responding disease (with no disease progression) after 4 courses may continue to receive study treatment for up to 1 year or discontinue study for alternative therapy at the discretion of the treating physician.

Patients are followed for survival.

PROJECTED ACCRUAL: A total of 13-26 patients will be accrued for this study within 1.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed Hodgkin's lymphoma* with any of the following histologies:

  * Not otherwise specified (NOS)
  * Mixed cellularity NOS
  * Lymphocytic depletion

    * NOS
    * Diffuse fibrosis
    * Reticular
  * Lymphocytic predominance

    * NOS
    * Diffuse
    * Nodular
  * Paragranuloma
  * Granuloma
  * Sarcoma
  * Nodular sclerosis

    * Cellular phase
    * NOS
    * Lymphocytic predominance
    * Mixed cellularity
    * Lymphocytic depletion NOTE: *Disease metastatic to bone marrow with granulocytopenia and/or thrombocytopenia is allowed, but is not evaluable for hematological toxicity
* Measurable disease by clinical or radiographic criteria
* Relapsed or refractory to conventional therapy

  * Received at least 2 prior cytotoxic chemotherapy regimens
* No stage IA or IIA nodal disease previously treated with any of the following:

  * Radiotherapy only
  * No more than 4 courses of prior chemotherapy

PATIENT CHARACTERISTICS:

Age

* 30 and under

Performance status

* Karnofsky 50-100% (over 16 years of age)
* Lansky 50-100% (16 and under) OR
* ECOG 0-2

Life expectancy

* At least 8 weeks

Hematopoietic

* See Disease Characteristics
* Absolute neutrophil count ≥ 750/mm^3
* Platelet count ≥ 75,000/mm^3 (transfusion independent, defined as ≥ 3 days since prior platelet transfusion)

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT ≤ 2.5 times ULN

Renal

* Creatinine clearance or radioisotope glomerular filtration rate ≥ 70 mL/min OR
* Creatinine based on age as follows:

  * No greater than 0.8 mg/dL (age 5 and under)
  * No greater than 1.0 mg/dL (age 6 to 10)
  * No greater than 1.2 mg/dL (age 11 to 15)
  * No greater than 1.5 mg/dL (over age 15)

Pulmonary

* DLCO ≥ 50%
* FEV_1 ≥ 50%
* Vital capacity ≥ 50%
* No evidence of dyspnea at rest
* No exercise intolerance

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study participation
* Seizure disorder allowed provided patient is on anticonvulsants and disorder is well controlled
* No evidence of active graft-versus-host disease

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Recovered from prior immunotherapy
* At least 6 months since prior allogeneic stem cell transplantation (SCT)
* At least 7 days since prior biologic agents
* More than 3 months since prior autologous SCT
* More than 1 week since prior growth factors
* No concurrent immunomodulating agents

Chemotherapy

* See Disease Characteristics
* More than 2 weeks since prior myelosuppressive chemotherapy (4 weeks for nitrosoureas) and recovered
* No prior gemcitabine and vinorelbine in combination (i.e., administered within 1 week of each other)

  * Prior gemcitabine or vinorelbine administered alone is allowed
* No other concurrent chemotherapy

Endocrine therapy

* No concurrent steroids, including corticosteroids as an antiemetic or for control of graft-versus-host disease

  * Concurrent corticosteroids allowed only for the following indications:

    * Adrenal crisis in patients with suppressed pituitary/adrenal response
    * Noncardiogenic pulmonary edema
    * Allergic reactions to amphotericin or transfusions treated with low-dose hydrocortisone (less than 100 mg/m^2)

Radiotherapy

* See Disease Characteristics
* At least 3 weeks since prior radiotherapy and recovered

Surgery

* Not specified

Other

* Concurrent immunosuppressive drugs allowed

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2004-07; Primary Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Tumor Response Rate | Up to 1 year
  Adequate tumor response is defined as achieving CR, VGPR or PR at any evaluation.

SECONDARY OUTCOMES:
Toxicities | Up to 4 weeks following the completion of therapy
  Toxic death, hepatic, cardiac or renal toxicity, hematologic toxicity, pulmonary toxicity or other grade 3 or 4 toxicities

CONTACTS AND LOCATIONS:
Overall Officials: Peter Cole, MD, Study Chair — Rutgers Cancer Institute of New Jersey
Locations (123):
- United States (108):
  - Lurleen Wallace Comprehensive Cancer at University of Alabama-Birmingham, Birmingham, Alabama
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Southern California Permanente Medical Group, Downey, California
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - Kaiser Permanente Medical Center - Oakland, Sacramento, California
  - Children's Hospital and Health Center - San Diego, San Diego, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Stanford Comprehensive Cancer Center - Stanford, Stanford, California
  - Carole and Ray Neag Comprehensive Cancer Center at the University of Connecticut Health Center, Farmington, Connecticut
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Lee Cancer Care of Lee Memorial Health System, Fort Myers, Florida
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Miami Children's Hospital, Miami, Florida
  - Florida Hospital Cancer Institute at Florida Hospital Orlando, Orlando, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - Sacred Heart Cancer Center at Sacred Heart Hospital, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - St. Joseph's Cancer Institute at St. Joseph's Hospital, Tampa, Florida
  - Kaplan Cancer Center at St. Mary's Medical Center, West Palm Beach, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Curtis & Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - St. Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Kosair Children's Hospital, Louisville, Kentucky
  - CancerCare of Maine at Eastern Maine Medial Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - Alvin and Lois Lapidus Cancer Institute at Sinai Hospital, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Floating Hospital for Children at Tufts - New England Medical Center, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - UMASS Memorial Cancer Center - University Campus, Worcester, Massachusetts
  - C.S. Mott Children's Hospital at University of Michigan Medical Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Spectrum Health Hospital - Butterworth Campus, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Breslin Cancer Center at Ingham Regional Medical Center, Lansing, Michigan
  - Children's Hospitals and Clinics of Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Medical Center & Children's Hospital - Fairview, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - Hackensack University Medical Center Cancer Center, Hackensack, New Jersey
  - St. Barnabas Medical Center Cancer Center, Livingston, New Jersey
  - Overlook Hospital, Morristown, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - University of New Mexico Cancer Research and Treatment Center, Albuquerque, New Mexico
  - Albany Medical Center Hospital, Albany, New York
  - Brooklyn Hospital Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Children's Medical Center - Dayton, Dayton, Ohio
  - Tod Children's Hospital, Youngstown, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Legacy Emanuel Hospital and Health Center & Children's Hospital, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Rhode Island Hospital Comprehensive Cancer Center, Providence, Rhode Island
  - Greenville Hospital System Cancer Center, Greenville, South Carolina
  - Sioux Valley Hospital and University of South Dakota Medical Center, Sioux Falls, South Dakota
  - T.C. Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Children's Hospital, Knoxville, Tennessee
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Texas Tech University Health Sciences Center School of Medicine - Amarillo, Amarillo, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - Baylor University Medical Center - Houston, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Providence Cancer Center at Sacred Heart Medical Center, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center - Tacoma, Tacoma, Washington
  - Madigan Army Medical Center - Tacoma, Tacoma, Washington
  - West Virginia University - Robert C. Byrd Health Sciences Center - Charleston Division, Charleston, West Virginia
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Princess Margaret Hospital for Children, Perth, Western Australia, Australia
- Canada (12):
  - University of Alberta Hospital, Edmonton, Alberta
  - CHUS-Hopital Fleurimont, Sherbrooke, Alberta
  - Children's & Women's Hospital of British Columbia, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Montreal Children's Hospital at McGill University Health Center, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec
  - Saskatoon Cancer Centre at the University of Saskatchewan, Saskatoon, Saskatchewan
  - Centre Hospitalier Universitaire de Quebec, Québec
- San Jorge Children's Hospital, Santurce, Puerto Rico
- Swiss Pediatric Oncology Group Geneva, Geneva, Switzerland

REFERENCES:
- [Result] Cole PD, McCarten KM, Drachtman RA, Alarcon Pd, Chen L, Trippett TM, Schwartz CL. Early [(1)(8)F]fluorodeoxyglucose positron emission tomography-based response evaluation after treatment with gemcitabine and vinorelbine for refractory Hodgkin disease: a children's oncology group report. Pediatr Hematol Oncol. 2010 Nov;27(8):650-7. doi: 10.3109/08880018.2010.504250. PMID 20863157
- [Result] Cole PD, Schwartz CL, Drachtman RA, de Alarcon PA, Chen L, Trippett TM. Phase II study of weekly gemcitabine and vinorelbine for children with recurrent or refractory Hodgkin's disease: a children's oncology group report. J Clin Oncol. 2009 Mar 20;27(9):1456-61. doi: 10.1200/JCO.2008.20.3778. Epub 2009 Feb 17. PMID 19224841